CLINICAL TRIAL: NCT02508389
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Trial of the Effects of GC4419 on Severe Oral Mucositis in Patients Receiving Cisplatin + Intensity-modulated Radiation Therapy (IMRT) for Locally Advanced Non-Metastatic Squamous Cell Carcinoma (SCC) of the Oral Cavity/Oropharynx
Brief Title: A Study of the Effects of GC4419 on Radiation Induced Oral Mucositis in Patients With Head/Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GT-201
Record Dates: First submitted 2015-07-16; First posted 2015-07-24 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Radiation Induced Oral Mucositis
Keywords: squamous cell carcinoma of the head and neck; oral cavity; oropharynx; intensity-modulated radiation therapy; chemotherapy; oral mucositis; superoxide dismutase; radioprotection
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Stomatitis | interventions — avasopasem manganese; Radiotherapy, Intensity-Modulated; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose GC4419: 30mg/day (Experimental): 30 mg GC4419/day prior to IMRT
  Interventions: Drug: Low Dose GC4419: 30mg/day; Radiation: Intensity-Modulated Radiation Therapy; Drug: Cisplatin
- High Dose GC4419: 90mg/day (Experimental): 90 mg GC4419/day prior to IMRT
  Interventions: Drug: High Dose GC4419: 90mg/day; Radiation: Intensity-Modulated Radiation Therapy; Drug: Cisplatin
- Placebo (Placebo Comparator): Placebo daily, prior to IMRT
  Interventions: Drug: Placebo; Radiation: Intensity-Modulated Radiation Therapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Low Dose GC4419: 30mg/day — Low Dose GC4419 will be administered by 60 minute IV infusion, within 1 hour prior to daily IMRT fractions, until IMRT is complete (generally M-F for approximately 7 weeks).
  Arms: Low Dose GC4419: 30mg/day
Drug: High Dose GC4419: 90mg/day — High Dose GC4419 will be administered by 60 minute IV infusion, within 1 hour prior to daily IMRT fractions, until IMRT is complete (generally M-F for approximately 7 weeks).
  Arms: High Dose GC4419: 90mg/day
Drug: Placebo — Placebo will be administered by 60 minute IV infusion, within 1 hour prior to daily IMRT fractions, until IMRT is complete (generally M-F for approximately 7 weeks).
  Arms: Placebo
Radiation: Intensity-Modulated Radiation Therapy — Daily fractions of IMRT (2.0-2.2 Gy) to a total of 60-72 Gy over approximately 7 weeks
Drug: Cisplatin — Administered 80-100 mg/m2 once every three weeks for 3 doses or 30-40 mg/m2 once weekly for 6-7 doses.
  Substitution of other systemic agents due to related toxicities (i.e., carboplatin) would be evaluated to determine eligibility by the Medical Monitor

SUMMARY:
The purpose of the phase 2, GT-201 clinical study is to determine if GC4419 administered prior to intensity-modulated radiation therapy (IMRT) reduces the incidence, duration, and severity of radiation induced oral mucositis in patients who have been diagnosed with locally advanced, non-metastatic squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
GT-201 is a randomized, double-blind, placebo-controlled, multi-center study conducted in the U.S. to evaluate GC4419 administered via an intravenous line (IV) for the reduction of incidence, duration, and severity of radiation induced oral mucositis in patients receiving cisplatin plus intensity-modulated radiation therapy for post-operative, or definitive treatment of locally advanced, non-metastatic squamous cell carcinoma of the head and neck, limited to the oral cavity or oropharynx. Patients will be randomized equally to 1 of 3 treatment arms:

Arm A: 30 mg GC4419 per day (60 min IV infusion to complete within 60 minutes prior to IMRT), concurrent with daily fractions of IMRT (2.0 - 2.2 Gy) to a total of 60 - 72 Gy over approximately 7 weeks, plus cisplatin administered 80 - 100 mg/m2 once every three weeks for 3 doses or 30 - 40 mg/m2 once weekly for 6-7 doses (investigator's choice).

Arm B: 90 mg GC4419 per day (60 min IV infusion to complete within 60 minutes prior to IMRT), concurrent with daily fractions of IMRT (2.0 - 2.2 Gy) to a total of 60 - 72 Gy over approximately 7 weeks, plus cisplatin administered 80 - 100 mg/m2 once every three weeks for 3 doses or 30 - 40 mg/m2 once weekly for 6-7 doses (investigator's choice).

Arm C: Placebo daily (60 min IV infusion to complete within 60 minutes prior to IMRT), concurrent with daily fractions of IMRT (2.0 - 2.2 Gy) to a total of 60 - 72 Gy over approximately 7 weeks, plus cisplatin administered 80 - 100 mg/m2 once every three weeks for 3 doses or 30 - 40 mg/m2 once weekly for 6-7 doses (investigator's choice).

Planned radiation fields in all 3 arms must include at least two oral sites (buccal mucosa, floor of mouth, tongue, soft palate) with each site receiving a dose of at least 50 Gy.

All patients will be assessed twice weekly for oral mucositis per WHO grading criteria until the completion of IMRT, and once weekly thereafter (if necessary) for 8 weeks, or until oral mucositis resolves to ≤ Grade 1.

Approximately 200 total to ensure that roughly 60 patients per arm receive study drug and complete requirements for primary endpoint analysis, which is defined as patients receiving a minimum cumulative dose of 60 Gy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically-confirmed diagnosis of squamous cell carcinoma of the head and neck, defined as SCC of the oral cavity or oropharynx that will be treated with cisplatin plus concurrent IMRT Note: Patients with unknown primary tumors whose treatment plan matches the requirements specified in Inclusion Criteria #2 and #3 below are eligible for the trial.
2. Treatment plan to receive a continuous course of IMRT delivered as single daily fractions of 2.0 to 2.2 Gy with a cumulative radiation dose between 60 Gy and 72 Gy. Planned radiation treatment fields must include at least two oral sites (buccal mucosa, floor of mouth, tongue, soft palate) that are each planned to receive a total of > 50 Gy. Patients who have had prior surgery are eligible, provided they have fully recovered from surgery, and patients who may have surgery in the future are eligible.
3. Treatment plan to receive standard cisplatin monotherapy administered either every three weeks (80-100 mg/m2 for 3 doses) or weekly (30-40 mg/m2 for 6-7 doses). The decision on which chemotherapy regimen to use in combination with IMRT and GC4419 will be at the discretion of the investigator.
4. Age 18 years or older
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
6. Adequate hematologic function as indicated by:

   * Absolute neutrophil counts (ANC) ≥ 1,500/mm3
   * Hemoglobin (Hgb) ≥ 9.0 g/dL
   * Platelet count ≥ 100,000/mm3
7. Adequate renal and liver function as indicated by:

   * Serum creatinine acceptable for treatment with cisplatin per institutional guidelines
   * Total bilirubin ≤ 1.5 x upper-normal limit (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
   * Alkaline phosphatase ≤ 2.5 x ULN
8. Human papilloma virus (HPV) status in tumor has been documented using tumor immunohistochemistry for HPV-p16 or other accepted test
9. Serum pregnancy test negative for females of childbearing potential
10. Males and females must agree to use effective contraception starting prior to the first day of treatment and continuing for 30 days after the last dose of GC4419
11. Properly obtained written informed consent

Exclusion Criteria:

1. Tumor of the lips, larynx, hypopharynx, nasopharynx, sinuses, or salivary glands
2. Metastatic disease (Stage IV C)
3. Prior radiotherapy to the region of the study cancer or adjacent anatomical sites or more than 25% of total body marrow-bearing area (potentially interfering with chemotolerance)
4. Prior induction chemotherapy
5. Receiving any approved or investigational anti-cancer agent other than those provided for in this study
6. Participation in another clinical trial or use of another investigational agent within 30 days of study entry
7. Requirement for significantly modified diet (liquids and/or solids) due to compromised oral/pharyngeal function at baseline
8. Requirement at baseline for parenteral or gastrointestinal tube-delivered nutrition for any reason
9. Malignant tumors other than head and neck cancer (HNC) within the last 5 years, unless treated definitively and with low risk of recurrence in the judgment of the treating investigator
10. Active infectious disease excluding oral candidiasis
11. Presence of oral mucositis (World Health Organization Score ≥ Grade 1) at study entry
12. Known history of HIV or active hepatitis B/C (patients who have been vaccinated for hepatitis B and do not have a history of infection are eligible)
13. Female patients who are pregnant or breastfeeding
14. Known allergies or intolerance to cisplatin and similar platinum-containing compounds
15. Requirement for concurrent treatment with nitrates or other drugs that may, in the judgment of the treating investigator, create a risk for a precipitous decrease in blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2015-10-12; Primary Completion 2017-09-18 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon T Holmlund, MD, Study Chair — Chief Medical Officer
Locations (64):
- United States (60):
  - University of Arizona Cancer Center at Dignity Health St. Joseph's, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences- Winthrop P. Rockefeller Cancer Institute, Little Rock, Arkansas
  - VA Long Beach Healthcare System, Long Beach, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Clinical Trials and Research Associates, Inc., Montebello, California
  - UC Irvine Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute, Stanford, California
  - St. Mary's Regional Cancer Center, Grand Junction, Colorado
  - UConn Health School of Dental Medicine, Farmington, Connecticut
  - Pasco Pinellas Cancer Center, Holiday, Florida
  - Lakeland Regional Health Cancer Center, Lakeland, Florida
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - Sacred Heart Medical Oncology Group, Pensacola, Florida
  - Northwestern University, Chicago, Illinois
  - University of Indianan, Goshen Center for Cancer Care, Goshen, Indiana
  - Department of Radiation Oncology University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Ashland-Bellefonte Cancer Center, Ashland, Kentucky
  - University of Kentucky, Albert B. Chandler Medical Center, Lexington, Kentucky
  - University of Louisville Hospital, James Graham Brown Cancer Center, Louisville, Kentucky
  - Tulane Cancer Center, New Orleans, Louisiana
  - CHRISTUS Schumpert Cancer Treatment Center, Shreveport, Louisiana
  - Baystate Regional Cancer Program, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Allegiance Health, Jackson, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Ellis Fichel Cancer Center, University of Missouri, Columbia, Missouri
  - Billings Clinic, Billings, Montana
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Renown Cancer Institute, Reno, Nevada
  - Hunterdon Hematology Oncology, LLC Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Jersey Shore University Medical Center- Hackensack Meridian Health, Neptune City, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - East Carolina University, Leo W. Jenkins Cancer Center, Greenville, North Carolina
  - Marion L. Shepard Cancer Center, Washington, North Carolina
  - Wake Forest Health, Winston-Salem, North Carolina
  - Ohio State University, James Cancer Center, Columbus, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - VA Portland Health Care System, Portland, Oregon
  - St. Luke's University Health Network, Easton, Pennsylvania
  - Thomas-Jefferson University Hospital-Bodine Center for Cancer Treatment, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Charleston Cancer Center, Charleston, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Prairie Lakes Health Care System, Watertown, South Dakota
  - Mountain States Health Alliance, Johnson City, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Texas Oncology, Plano, Texas
  - Scott and White Memorial Hospital and Clinic, Temple, Texas
  - Hope Cancer Center, Tyler, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - Providence Regional Medical Center, Everett, Washington
  - VA Puget Sound Health Care System, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
- Canada (3):
  - Northeast Cancer Centre, Health Sciences North, Greater Sudbury, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Centre intégré universitaire de santé et de services sociaux de la Mauricie-et-du-centre-du-Québec, Trois-Rivières, Quebec
- Fundación de Investigación, San Juan, PR, Puerto Rico

REFERENCES:
- [Derived] Mapuskar KA, Vasquez Martinez G, Pulliam CF, Petronek MS, Steinbach EJ, Monga V, Furqan M, Jetton JG, Saunders DP, Pearce A, Davidson S, Pitre L, Dunlap NE, Fairbanks R, Lee CM, Mott SL, Bodeker KL, Cl H, Buatti JM, Anderson CM, Beardsley RA, Holmlund JT, Zepeda-Orozco D, Spitz DR, Allen BG. Avasopasem manganese (GC4419) protects against cisplatin-induced chronic kidney disease: An exploratory analysis of renal metrics from a randomized phase 2b clinical trial in head and neck cancer patients. Redox Biol. 2023 Apr;60:102599. doi: 10.1016/j.redox.2022.102599. Epub 2023 Jan 3. PMID 36640725
- [Derived] Anderson CM, Lee CM, Saunders D, Curtis AE, Dunlap NE, Nangia C, Lee AS, Kovoor P, Bar-Ad V, Pedadda AV Jr, Holmlund J, Downs M, Sonis ST. Two-Year Tumor Outcomes of a Phase 2B, Randomized, Double-Blind Trial of Avasopasem Manganese (GC4419) Versus Placebo to Reduce Severe Oral Mucositis Owing to Concurrent Radiation Therapy and Cisplatin for Head and Neck Cancer. Int J Radiat Oncol Biol Phys. 2022 Nov 1;114(3):416-421. doi: 10.1016/j.ijrobp.2022.06.063. Epub 2022 Jun 17. PMID 35724774

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose GC4419: 30mg/Day: 30 mg GC4419/day prior to IMRT
  Low Dose GC4419: 30mg/day: Low Dose GC4419 will be administered by 60 minute IV infusion, within 1 hour prior to daily IMRT fractions, until IMRT is complete (generally M-F for approximately 7 weeks).
  Intensity-Modulated Radiation Therapy: Daily fractions of IMRT (2.0-2.2 Gy) to a total of 60-72 Gy over approximately 7 weeks
  Cisplatin: Administered 80-100 mg/m2 once every three weeks for 3 doses or 30-40 mg/m2 once weekly for 6-7 doses.
  Substitution of other systemic agents due to related toxicities (i.e., carboplatin) would be evaluated to determine eligibility by the Medical Monitor
- High Dose GC4419: 90mg/Day: 90 mg GC4419/day prior to IMRT
  High Dose GC4419: 90mg/day: High Dose GC4419 will be administered by 60 minute IV infusion, within 1 hour prior to daily IMRT fractions, until IMRT is complete (generally M-F for approximately 7 weeks).
  Intensity-Modulated Radiation Therapy: Daily fractions of IMRT (2.0-2.2 Gy) to a total of 60-72 Gy over approximately 7 weeks
  Cisplatin: Administered 80-100 mg/m2 once every three weeks for 3 doses or 30-40 mg/m2 once weekly for 6-7 doses.
  Substitution of other systemic agents due to related toxicities (i.e., carboplatin) would be evaluated to determine eligibility by the Medical Monitor
- Placebo: Placebo daily, prior to IMRT
  Placebo: Placebo will be administered by 60 minute IV infusion, within 1 hour prior to daily IMRT fractions, until IMRT is complete (generally M-F for approximately 7 weeks).
  Intensity-Modulated Radiation Therapy: Daily fractions of IMRT (2.0-2.2 Gy) to a total of 60-72 Gy over approximately 7 weeks
  Cisplatin: Administered 80-100 mg/m2 once every three weeks for 3 doses or 30-40 mg/m2 once weekly for 6-7 doses.
  Substitution of other systemic agents due to related toxicities (i.e., carboplatin) would be evaluated to determine eligibility by the Medical Monitor
Period: Overall Study
Arm/Group | Low Dose GC4419: 30mg/Day | High Dose GC4419: 90mg/Day | Placebo
Started | 73 | 76 | 74
Completed | 45 | 45 | 42
Not Completed | 28 | 31 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose GC4419: 30mg/Day | High Dose GC4419: 90mg/Day | Placebo | Total
Number analyzed (Participants) | 73 | 76 | 74 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (9.10) | 57.6 (10.6) | 57.9 (9.61) | 57.7 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 10 | 31
  Male | 64 | 64 | 64 | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 2 | 8
  Not Hispanic or Latino | 68 | 72 | 70 | 210
  Unknown or Not Reported | 3 | 0 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 4 | 10
  White | 69 | 71 | 68 | 208
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Duration (in Days) of Radiation Induced Severe Oral Mucositis (OM) Per World Health Organization (WHO) Criteria
Description: Assessed from the first determination of ≥Grade 3 OM to the first instance of non-severe OM (≤Grade 2), without a subsequent instance of ≥Grade 3
Time Frame: From start of Intensity-modulated radiation therapy (IMRT) through 8 weeks follow-up, an average of 15 weeks
Population: intent to treat population
Measure: Median (Full Range); unit: days
Arm/Group | Low Dose GC4419: 30mg/Day | High Dose GC4419: 90mg/Day | Placebo
Number analyzed (Participants) | 73 | 76 | 74
days | 8 [0 to 93] | 1.5 [0 to 100] | 19 [0 to 83]

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Number of participants with treatment emergent adverse events (TEAE) per arm
Time Frame: First dose of IMRT through the completion of IMRT, estimated to be up to 7 weeks.
Population: Treated Population
Measure: Number; unit: participants
Arm/Group | Low Dose GC4419: 30mg/Day | High Dose GC4419: 90mg/Day | Placebo
Number analyzed (Participants) | 73 | 72 | 72
participants
  Number of Subjects with at least one TEAE | 73 | 72 | 72
  Number of Subjects with at least one serious TEAE | 34 | 34 | 28

3. Secondary Outcome: Number of Participants Who Experience Severe OM
Description: Number of participants who experience severe OM from the first IMRT fraction through the last IMRT fraction
Time Frame: Minimum of 60 Gy administered to tumor, approximately 30 IMRT fractions, which is estimated to be 6-7 weeks.
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Low Dose GC4419: 30mg/Day | High Dose GC4419: 90mg/Day | Placebo
Number analyzed (Participants) | 73 | 76 | 74
participants | 29 | 28 | 43

4. Secondary Outcome: Number of Participants Who Experienced Grade 4 OM From the First IMRT Fraction Through the Last IMRT Fraction
Description: Number of Participants who experienced Grade 4 OM
Time Frame: First dose of IMRT through the completion of IMRT, estimated to be up to 6-7 weeks.
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Low Dose GC4419: 30mg/Day | High Dose GC4419: 90mg/Day | Placebo
Number analyzed (Participants) | 73 | 76 | 74
participants | 44 | 33 | 48

5. Secondary Outcome: Number of IMRT Fractions Delivered at Onset of Severe OM
Description: Onset of severe OM: number of IMRT fractions delivered at onset of severe OM
Time Frame: Onset of Severe OM, estimated to be between first dose of IMRT and 7 weeks.
Population: Intent to treat population
Measure: Median (95% Confidence Interval); unit: IMRT Fractions
Arm/Group | Low Dose GC4419: 30mg/Day | High Dose GC4419: 90mg/Day | Placebo
Number analyzed (Participants) | 73 | 76 | 74
IMRT Fractions | 33 [25.00 to 35.00] | 35 [28.00 to 35.00] | 28 [22.00 to 33.00]

6. Secondary Outcome: Number of Participants Who Experienced Grade 4 Oral Mucocitis (OM) From the First IMRT Fraction Through the Last IMRT Fraction
Description: Number of Participants who experienced Grade 4 OM
Time Frame: Onset of Grade 4 OM, estimated to be between first dose of IMRT and 7 weeks.
Population: Intent to Treat Population
Measure: Number; unit: participants
Arm/Group | Low Dose GC4419: 30mg/Day | High Dose GC4419: 90mg/Day | Placebo
Number analyzed (Participants) | 73 | 76 | 74
participants | 15 | 12 | 22

7. Secondary Outcome: Number of Participants With Tumor Outcomes Defined as Locoregional Failure, Distant Metastases, Disease Progression and Deaths
Description: Effect of treatment assignment on tumor outcomes (locoregional failure, distant metastases, progression-free survival, overall survival) Only 73 subjects in Placebo Arm were analyzed for locoregional failure, distant disease and progression-free survival because 1 subject was determined after enrollment to have a non-head and neck cancer and was therefore excluded from these analyses
Time Frame: Up to 1 year following completion of chemoradiation.
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose GC4419: 30mg/Day | High Dose GC4419: 90mg/Day | Placebo
Number analyzed (Participants) | 73 | 76 | 74
Participants
  Number With Locoregional Failure: number analyzed (Participants) | 73 | 76 | 73
  Number With Locoregional Failure | 7 | 6 | 5
  Number With Distant Disease: number analyzed (Participants) | 73 | 76 | 73
  Number With Distant Disease | 9 | 6 | 6
  Number with Progressive Disease: number analyzed (Participants) | 73 | 76 | 73
  Number with Progressive Disease | 15 | 12 | 11
  Number of Deaths | 11 | 10 | 10

ADVERSE EVENTS:
Time Frame: from first dose study drug through 30 days after last dose, approximately 11 weeks
Description: All-cause mortality was reported for all randomized intent-to-treat subjects (ITT) (inclusive of randomization failures who did not get treated). Adverse Events (AEs)/Serious Adverse Events (SAEs) were analyzed for only subjects who received at least one dose of study drug (treated population)
Arm/Group | Low Dose GC4419: 30mg/Day | High Dose GC4419: 90mg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 1/73 | 1/76 | 2/73
Serious Adverse Events (participants affected / at risk) | 34/73 | 34/72 | 28/72
Other Adverse Events (participants affected / at risk) | 73/73 | 72/72 | 72/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose GC4419: 30mg/Day (N=73) | High Dose GC4419: 90mg/Day (N=72) | Placebo (N=72)
Lung Infection (Infections and infestations) | 1 | 2 | 2
Pneumonia (Infections and infestations) | 0 | 2 | 3
Sepsis (Infections and infestations) | 1 | 1 | 2
Clostridium difficile infection (Infections and infestations) | 2 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Cellulitis streptococcal (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 6
Nausea (Gastrointestinal disorders) | 3 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Dehydration (Gastrointestinal disorders) | 1 | 3 | 2
Decreased appetite (Gastrointestinal disorders) | 0 | 0 | 3
Hyponatraemia (Gastrointestinal disorders) | 2 | 1 | 0
Malnutrition (Gastrointestinal disorders) | 1 | 2 | 0
Failure to thrive (Gastrointestinal disorders) | 2 | 0 | 0
Hyperglycaemia (Gastrointestinal disorders) | 1 | 0 | 0
Hypocalcaemia (Gastrointestinal disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 4 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 3 | 2
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 4 | 1
Pyrexia (General disorders) | 3 | 2 | 0
Asthenia (General disorders) | 1 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Atrial flutter (Cardiac disorders) | 2 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose GC4419: 30mg/Day (N=73) | High Dose GC4419: 90mg/Day (N=72) | Placebo (N=72)
Nausea (Gastrointestinal disorders) | 50 | 59 | 54
Constipation (Gastrointestinal disorders) | 43 | 46 | 38
Vomiting (Gastrointestinal disorders) | 38 | 35 | 34
Dysphagia (Gastrointestinal disorders) | 31 | 34 | 31
Diarrhoea (Gastrointestinal disorders) | 31 | 22 | 28
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 12 | 11
Dyspepsia (Gastrointestinal disorders) | 13 | 8 | 6
Salivary hypersecretion (Gastrointestinal disorders) | 6 | 11 | 3
Odynophagia (Gastrointestinal disorders) | 6 | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 4
Glossodynia (Gastrointestinal disorders) | 3 | 4 | 1
Lymphopenia (Blood and lymphatic system disorders) | 67 | 63 | 64
Leukopenia (Blood and lymphatic system disorders) | 27 | 28 | 28
Neutropenia (Blood and lymphatic system disorders) | 18 | 17 | 19
Anaemia (Blood and lymphatic system disorders) | 20 | 17 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 7 | 10
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 6 | 3
Cytopenia (Blood and lymphatic system disorders) | 5 | 1 | 2
Fatigue (General disorders) | 44 | 47 | 50
Pyrexia (General disorders) | 15 | 13 | 15
Chills (General disorders) | 10 | 11 | 10
Oedema peripheral (General disorders) | 5 | 8 | 6
Asthenia (General disorders) | 3 | 4 | 5
Face oedema (General disorders) | 3 | 3 | 4
Pain (General disorders) | 1 | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 27 | 30 | 23
Decreased appetite (Metabolism and nutrition disorders) | 22 | 31 | 23
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 21 | 13
Hypomagnesaemia (Metabolism and nutrition disorders) | 16 | 18 | 16
Hyponatraemia (Metabolism and nutrition disorders) | 11 | 7 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 5 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 3 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 5 | 3
Malnutrition (Metabolism and nutrition disorders) | 2 | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 46 | 44 | 46
Hiccups (Respiratory, thoracic and mediastinal disorders) | 17 | 19 | 17
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 16 | 16 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 8 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 8
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 7
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2
Dysgeusia (Nervous system disorders) | 40 | 31 | 35
Headache (Nervous system disorders) | 16 | 24 | 17
Dizziness (Nervous system disorders) | 16 | 19 | 9
Paraesthesia (Nervous system disorders) | 7 | 12 | 9
Syncope (Nervous system disorders) | 4 | 5 | 4
Oral candidiasis (Infections and infestations) | 33 | 31 | 21
Candida infection (Infections and infestations) | 13 | 11 | 12
Urinary tract infection (Infections and infestations) | 4 | 6 | 2
Mucosal infection (Infections and infestations) | 5 | 2 | 3
Stoma site infection (Infections and infestations) | 0 | 5 | 3
Radiation skin injury (Injury, poisoning and procedural complications) | 37 | 38 | 34
Stoma site pain (Injury, poisoning and procedural complications) | 8 | 1 | 6
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 4
Weight decreased (Investigations) | 29 | 32 | 25
Electrocardiogram QT prolonged (Investigations) | 6 | 5 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 12 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 7 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 9 | 3
Erythema (Skin and subcutaneous tissue disorders) | 1 | 4 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 5 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 | 4 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 0 | 3
Hypotension (Vascular disorders) | 12 | 17 | 7
Hypertension (Vascular disorders) | 7 | 12 | 10
Flushing (Vascular disorders) | 8 | 2 | 2
Orthostatic hypotension (Vascular disorders) | 4 | 2 | 4
Deep vein thrombosis (Vascular disorders) | 4 | 1 | 3
Tinnitus (Ear and labyrinth disorders) | 19 | 15 | 19
Ear pain (Ear and labyrinth disorders) | 5 | 5 | 4
Hearing impaired (Ear and labyrinth disorders) | 6 | 2 | 4
Insomnia (Psychiatric disorders) | 11 | 11 | 8
Anxiety (Psychiatric disorders) | 8 | 6 | 7
Depression (Psychiatric disorders) | 1 | 4 | 6
Confusional state (Psychiatric disorders) | 0 | 4 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 9 | 7
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 3 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2
Acute kidney injury (Renal and urinary disorders) | 10 | 5 | 8
Renal disorder (Renal and urinary disorders) | 4 | 5 | 4
Sinus tachycardia (Cardiac disorders) | 2 | 4 | 0
Vision blurred (Eye disorders) | 0 | 7 | 2
Flatulence (Gastrointestinal disorders) | 0 | 5 | 0
Pharyngitis (Infections and infestations) | 1 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT02508389/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT02508389/SAP_001.pdf